CLINICAL TRIAL: NCT07360405
Title: Diet-Based Treatment for Migraine Relief
Brief Title: Dietary Intervention for Migraine Relief
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Principal Investigator, Kathleen Holton, Professor, American University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-297
Record Dates: First submitted 2025-12-19; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Migraine; Chronic pain; Diet; Glutamate
MeSH Terms: conditions — Migraine Disorders; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Parallel-arm design followed by a crossover, double-blind, placebo-controlled challenge with monosodium glutamate (MSG) versus placebo.
Masking Description: Masking is not possible in this trial as the nature of intervention is diet based.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet group (Active Comparator)
  Interventions: Behavioral: Dietary training
- Control group (No Intervention): This group will follow their own diet without any intervention. However after this period, they will given the chance of receiving intervention as well.

INTERVENTIONS:
Behavioral: Dietary training — Subjects will undergo a 2-hour online training session to teach them how to follow the low glutamate diet. The low glutamate diet is a healthy, whole-food diet designed to limit the intake of free glutamate/aspartate, while also emphasizing the consumption of foods which are high in nutrients that protect against glutamate excitotoxicity and oxidative stress.
  Other Names: Low glutamate diet
  Arms: Diet group

SUMMARY:
The goal of this clinical trial is to evaluate whether a low-glutamate diet can improve migraine symptoms in adults with migraine and to explore possible biological changes associated with dietary improvement. The study focuses on whether reducing dietary glutamate intake may influence processes involved in migraine, such as brain excitation, inflammation, and oxidative stress.

The main questions this study aims to answer are:

Does following a low-glutamate diet reduce the number of migraine days and the severity and duration of migraine attacks, and improve quality of life?

Are improvements in migraine symptoms associated with changes in blood-based biological markers related to migraine activity?

Researchers will compare participants assigned to the low-glutamate diet with participants assigned to a wait-list control group to evaluate differences in migraine outcomes and related biological measures.

Participants will:

Complete a baseline run-in period while tracking headaches using a daily migraine diary

Either follow a low-glutamate dietary intervention or continue their usual diet as part of a wait-list control

Complete standardized questionnaires related to migraine symptoms and quality of life

Provide blood samples for laboratory analyses

Undergo neuroimaging assessments (for a subset of participants)

DETAILED DESCRIPTION:
The purpose of this clinical trial is to evaluate whether a low-glutamate diet is an effective treatment for migraine and to explore how this dietary approach may influence biological processes related to migraine. The low-glutamate diet reduces intake of free glutamate commonly found in ultra-processed foods and food additives, while emphasizing whole foods rich in nutrients that support brain health and reduce oxidative stress.

The study is based on prior research showing that this diet led to substantial improvements in migraine symptoms among individuals with chronic pain, with migraine remission often observed after one month. These improvements were also associated with measurable changes in brain structure, suggesting a potential link between dietary glutamate exposure and migraine-related brain changes.

The primary goals of this study are to:

Determine whether one month on a low-glutamate diet reduces migraine frequency, severity, and duration and improves quality of life

Examine changes in blood markers related to migraine pain signaling

Assess whether dietary changes are associated with changes in brain structure or chemistry in a subset of participants

Participants will first complete a 4-week run-in period during which they will continue their usual diet and record headaches and migraines using a daily electronic diary. Eligible participants will then be randomly assigned to either begin the low-glutamate diet immediately or continue their usual diet for one additional month (wait-list control). All participants will complete questionnaires, provide blood and urine samples, and undergo in-person assessments at the end of each study phase. A subset of participants will also undergo Magnetic Resonance Imaging (MRI) scans.

Participants assigned to the diet will receive structured dietary training, educational materials, and weekly follow-up support to promote adherence. After the initial dietary phase, participants will complete a double-blind, placebo-controlled crossover challenge, during which they will receive short courses of monosodium glutamate (MSG) and placebo while remaining on the low-glutamate diet. This phase is designed to determine whether migraine symptoms return specifically in response to glutamate exposure.

Throughout the study, participants will continue to track migraine symptoms using daily diaries. The results of this study may help determine whether a low-glutamate diet is a safe, non-pharmacologic treatment option for migraine and may provide insight into dietary factors that contribute to migraine development and persistence.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all races and ethnicities
* Age 18-75 years
* Documented diagnosis of chronic or episodic migraine for at least 6 months, based on International Classification of Headache Disorders, 3rd edition (ICHD-III) criteria, defined as:

  * 8 headache days per month, and
  * 4 migraine days per month
* Migraine onset before age 50
* On a stable medication regimen for at least 1 month prior to enrollment
* Willing to maintain stable medications throughout the study
* Willing to discontinue supplements during the study period
* Women of childbearing potential must be willing to use birth control during the study timeframe

Exclusion Criteria:

* Current pregnancy, plans to become pregnant during the study timeframe, or current breastfeeding
* Current use of medications affecting glutamatergic or gamma-Aminobutyric Acid (GABA) neurotransmission (unless discontinued under physician guidance)
* Current use of quarterly injectable migraine preventive medications
* Unwillingness to modify dietary intake or to stop alcohol and marijuana use during the study
* Substance use disorder within the past year
* Diagnosed seizure disorder
* Severe asthma requiring past hospitalization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Migraine days | 4 weeks
  Changes in the number of migraine days with improvement defined as a ≥50% reduction in migraine days
Patient Global Impression of Change | 4 weeks
  Changes in the patient Global Impression of Change score, where in this study improvement defined as the score of "much" or "very much" improved. This measure is a simple 1-to-7 scale where patients rate how much their condition or symptoms have improved. 1 means very much improved and 7 means very much worse.

SECONDARY OUTCOMES:
Migraine-specific quality of life | 4 weeks
  Changes in the quality of life measured by the migraine-specific quality of life. This questionnaire scored 0-100 (higher is better).
Migraine duration | 4 weeks
  Change in migraine duration (hours)
Migraine intensity | 4 weeks
  Change in migraine intensity, measured in scale of 0 (least pain) to 10 (highest pain).
Skin carotenoid levels | 4 weeks
  Change in the skin carotenoid levels (the score is measured by a biophotonic scanner)
Skin carotenoid levels | 4 weeks
  Change in Skin carotenoid levels being measure using a biophotonic scanner
Glutathione | 4 weeks
  Change in the blood levels of glutathione (micromol/L)
Coenzyme Q10 | 4 weeks
  Change in the serum level of coenzyme Q10 (mcg/mL)
8-hydroxydeoxyguanosine (8OHdG) | 4 weeks
  Change in the urine levels of 8-hydroxydeoxyguanosine (8OHdG) (mcg/g Creatinine)
Lipid peroxides | 4 weeks
  Change in the urine level of lipid peroxides (micromol/g Creatinine)
Glutamate | 4 weeks
  Change in the plasma levels of glutamate (micromol/dL)
Aspartate | 4 weeks
  Change in the plasma levels of aspartate (micromol/dL)
Calcitonin gene-related peptide (CGRP) | 4 weeks
  Change in the serum calcitonin gene-related peptide (CGRP) level
Brain levels of glutamate | 4 weeks
  Measuring the change in the level of glutamate in brain using Magnetic resonance spectroscopy (MRS)
Brain level of glutathione | 4 weeks
  Measuring the change in the level of glutathione in brain using Magnetic resonance spectroscopy (MRS)
Visual cortex thickness | 4 weeks
  Changes in the visual cortex thickness measured via Magnetic Resonance Imaging (MRI)
Blood brain barrier permeability | 4 weeks
  Change in blood brain barrier permeability will be assessed using magnetic resonance imaging (MRI) with 3-dimensional diffusion-prepared arterial spin labeling (3D DP-ASL), a non-invasive imaging technique for quantifying blood-brain barrier permeability.

CONTACTS AND LOCATIONS:
Locations (1):
- American University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No